CLINICAL TRIAL: NCT00929890
Title: Effect of Weight Loss Through Dietary Energy Restriction With or Without Exercise on Vascular and Metabolic Parameters in Subjects With Obesity
Brief Title: Additional Metabolic and Vascular Effects of Exercise in Patients on Diet-based Weight Loss Programs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 08282
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-07

CONDITIONS: Obesity
Keywords: Obesity; Exercise; Diet; Lifestyle; Vascular reactivity; Body composition; Lipids; Glucose; Insulin resistance
MeSH Terms: conditions — Obesity; Motor Activity; Insulin Resistance | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling (Active Comparator): Patients will receive dietary counseling and a general advice on physical activity
  Interventions: Behavioral: General lifestyle, diet and physical activity counselling
- Exercise training (Experimental): patients will receive dietary counseling and will be enrolled in supervised exercise training
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: General lifestyle, diet and physical activity counselling — Low-calorie, balanced diet and a general advice on the importance of regular physical activity
  Arms: Lifestyle counseling
Behavioral: Exercise training — Subject will receive dietary counselling (low-calorie, balanced diet) and will be enrolled in a supervised, 3 times a week, exercise training program
  Arms: Exercise training

SUMMARY:
This study tests the hypothesis that exercise training can confer additional benefit to patients in weight-loss programs in the form of improvements in either metabolic or vascular parameters or both. Patients will be randomized to either diet plus conventional physical activity or diet plus a planned exercise training. The interventions will be carried out until the patients lose between 5% and 7.5% of their initial weight. At entry and at the end, all subjects will be evaluated for outcomes such as blood glucose, lipid profile, insulin, c-reactive protein, fibrinogen, vascular reactivity (doppler ultrasound) and total and abdominal visceral fat (CT-scan). Both groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* BMI> 30 and <40

Exclusion Criteria:

* Diabetes mellitus
* Active endocrine disease
* Active heart disease
* Active smoking
* Medical contra-indications for exercise
* Using anti-obesity drugs

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-02; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Reduction in homeostasis model assessment of insulin resistance (HOMA-IR) | 6 months
Change in lipid profile | 6 months
Reduction in abdominal (visceral) fat | 6 months
Change in vascular reactivity | 6 months

SECONDARY OUTCOMES:
C-reactive protein | 6 months
Fibrinogen | 6 months
vonWillebrand factor | 6 months
Waist circumference | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rogério Friedman, MD, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre, Universidade Federal do Rio Grande do Sul
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Lopes AL, Macedo RCO, Kruger RL, Friedman R, Carteri RB, Reischak-Oliveira A. Fasted exercise does not improve postprandial lipemia responses to different meals in lean and obese subjects: A crossover, randomized clinical trial. Clin Nutr ESPEN. 2021 Feb;41:160-167. doi: 10.1016/j.clnesp.2020.11.013. Epub 2020 Dec 30. PMID 33487260